CLINICAL TRIAL: NCT00918684
Title: Aging White Matter Changes, Executive Dysfunction and Depression
Brief Title: Aging Brain Changes, Executive Dysfunction and Depression
Acronym: FA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0204005523; R01MH065653-01A1 (NIH)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): 12-week open label with 2 week placebo period (14 weeks total)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10mg tab daily
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to look at the relationship between age related structural brain changes and changes in depressive symptoms,disability and several aspects of cognitive functioning following treatment with escitalopram.

DETAILED DESCRIPTION:
Age-related brain changes have been associated with development of late-life depression. Prominent among aging-related changes is decline in white matter disproportionately affecting frontal structures.Based on previous findings, we conceptualized treatment resistance, disability, and executive dysfunction as clinical phenomena contributed, at least in part, by compromised integrity of frontal neural systems. The study focuses on frontal white matter abnormalities in geriatric depression and their relationship to treatment response, disability,and executive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Two strata: 60-74 years (n=60) subjects and 75-84 years (n=60).
2. Diagnosis: Major depression, unipolar (by DSM-IV criteria); or, for control subjects, no diagnosis of major depression, no history of depression or other psychiatric conditions.
3. Severity of depression: A 24-Item HDRS above 19; Level of Executive Dysfunction: Two strata within each age stratum: Stroop Color-Word scores below and above 24 (1 SD below the median of our normal elderly sample).

Exclusion Criteria:

1. Psychotic depression by DSM-IV, i.e., presence of delusions with a score higher than 2 (questionable delusion) rated by the Scale for Assessment of Positive Symptoms (SAPS; 51).
2. High suicide risk, i.e. intent or plan to attempt suicide in near future.
3. Presence of any Axis I psychiatric disorder or substance abuse other than unipolar major depression.
4. Axis II diagnosis of antisocial personality (by SCID-P and DSM-IV).
5. History of psychiatric disorders other than unipolar major depression or generalized anxiety disorder (bipolar disorder, hypomania, are exclusion criteria).
6. Cognition: MMSE scores below 24 or diagnosis of dementia by DSM-IV.
7. Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs known to cause depression, e.g., reserpine, alpha-methyl-dopa, steroids.
8. Failure to respond to an adequate trial of escitalopram (10 mg/day or more for 6 weeks or longer) during the current or previous depressive episodes.
9. Current involvement in psychotherapy.
10. History of hypersensitivity to escitalopram or need to receive drugs that may interact with escitalopram.
11. Inability to perform any of the ADLs (MAI: ADL subscale) even with assistance, e.g. walking with a cane is not an exclusion criterion.
12. Inability to speak English.
13. Aphasia.
14. Residence outside a 45-minute drive from Cornell's clinical facilities.
15. Patients taking MAOI's and Fluoxetine will be excluded.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2002-12 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow of the Overall Study
Pre-assignment Details: 116 participants were consented and enrolled. 10 of these subjects did not participate in the washout/placebo phase.
Period: Two Week Drug Washout and Placebo Phase
Arm/Group | Escitalopram
Started | 106
Completed | 90
Not Completed | 16
Not completed — Placebo Reponder | 16
Period: Treatment Phase
Arm/Group | Escitalopram
Started | 90
Completed | 65
Not Completed | 25
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 8
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: All subjects who entered the treatment phase
Arm/Group | Escitalopram
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.82 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90
Hamilton Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Scale for Depression 24 item total scores range from 0-76. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
  units on a scale | 21.21 (4.51)
Mini Mental Status Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — MMSE total scores range from 0-30. Higher scores indicate better memory functioning (no cognitive impairment). Total scores are reported with no subscales.
  units on a scale | 28.08 (1.64)
WHODAS-II Disability Score [Mean (Standard Deviation); unit: units on a scale] — WHODAS II total scores can range from 0-100. Higher scores indicate greater severity of disability. Total scores are reported with no subscales.
  units on a scale | 34.64 (10.56)
Stroop Color-Word Test [Mean (Standard Deviation); unit: units on a scale] — Stroop Color-Word total scores can range from 0-100. Higher scores indicate better memory functioning (no cognitive impairment). Total scores are reported with no subscales.
  units on a scale | 32.77 (10.63)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale.
Description: A published and widely-used scale for rating depression severity, the Hamilton Depression Rating Scale 24 item total scores range from 0-76. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
Time Frame: 14 weeks (12th week of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 90
units on a scale | 8.09 (5.93)

2. Primary Outcome: WHODAS-II Disability Scale
Description: A disability rating scale published by the World Health Organization, the WHODAS II total scores can range from 0-100. Higher scores indicate greater severity of disability. Total scores are reported with no subscales.
Time Frame: 14 weeks (12th week of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 90
units on a scale | 31.43 (9.14)

3. Primary Outcome: Stroop Color-Word Test
Description: A published and widely used executive dysfunction test, the Stroop Color-Word total scores can range from 0-100. Higher scores indicate better memory functioning (no cognitive impairment). Total scores are reported with no subscales.
Time Frame: 14 weeks (12th week of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 90
units on a scale | 33.63 (10.2)

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Description: Clinicaltrials.gov definitions apply.
Arm/Group | Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 6/90
Other Adverse Events (participants affected / at risk) | 55/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=90)
Non-cardiac chest pain (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=90)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anorgasmia (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Prolonged bleeding after a cut (Blood and lymphatic system disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (15)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Prolonged gum bleeding (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Vascular disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Homicidal ideation (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Reproductive system and breast disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No